CLINICAL TRIAL: NCT06106555
Title: Vilka Faktorer påverkar Behandlingsutfall Vid Dialektisk Beteendeterapi för Borderline Personlighetssyndrom?
Brief Title: Which Factors Are Relevant for Treatment Outcome in Dialectical Behaviour Therapy for Borderline Personality Disorder?
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Department of Psychology. Lund University. (Unknown); University of Toronto (Other); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Dnr 2023-03990-01
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Borderline Personality Disorder; Non-suicidal Self-injury; Deliberate Self Harm
Keywords: Borderline Personality Disorder; Dialectical Behavior Therapy; Deliberate Self-Harm; Non-suicidal Self-injury; Self-concept; Personality
MeSH Terms: conditions — Borderline Personality Disorder; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with BPD: Individuals with BPD, as defined by the DSM-V, and a recent history (past 12 months) of self-harming behaviour.
  Interventions: Behavioral: Dialectibal Behaviour Therapy

INTERVENTIONS:
Behavioral: Dialectibal Behaviour Therapy — Standard Dialectical Behaviour Therapy of up to 12 months as described Professor Linehan

SUMMARY:
The objective of this project is to investigate factors that contribute to the success and lack of success in DBT among individuals with BPD and a history of self-harm in a clinical psychiatric setting.

1. Do certain personality factors and identity disturbance predict the treatment outcome of DBT in individuals with BPD?
2. Do changes in identity disturbance, self-hate, or emotion regulation mediate the treatment outcome of DBT in individuals with BPD?
3. Do specific personality profiles moderate the treatment outcomes of DBT for individuals with BPD?
4. When does the primary treatment effect occur, and does this effect persist after a 12-month follow-up period?

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a complex and enduring mental health condition characterized by a range of symptoms. The consequences of BPD are severe, causing individual suffering, impairments in daily functioning, and increased mortality rates. Dialectical behavior therapy (DBT) is one of the most widely used treatment models for BPD and self-harm. DBT has demonstrated positive outcomes but not all individuals benefit equally from this therapy, highlighting the need for further exploration. Specifically, there is a knowledge gap regarding what predicts positive treatment response. Research exploring this topic, has highlighted the potential significance of emotion regulation, personality profiles, self-concept, and identity disturbance in understanding the outcomes of individuals with BPD.

The primary objective of this research project is to investigate the factors that contribute to the success and lack of success in DBT.

All individuals referred to DBT-treatment in the Adult psychiatric clinic in Lund will be offered participation in the study. All study participants receive the same treatment as those who chose not to participate. Measures will commence after treatment contracts have been negotiated and the treatment will continue up to a maximum treatment length of one year.

Data will be retrieved from databases, medical records as well as collected as self-report forms. Self-report measures will be conducted every three months, at end of treatment and at follow up 12 months after end of treatment. Data from registries and charts will be collected at time of consent and at follow up 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Borderline personality disorder as defined by the DSM-V (assessed with SCID or uquivalent).
* Self-harm over the past 12 months
* Offered DBT at the Lund adult psychiatric clinic

Exclusion Criteria:

* Unable to read or communicate in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Borderline personality disorder in a specialized psychiatric setting. A majority of the individuals will have comorbid psychiatric conditions and have been offered other pharmacological and psychological treatments through their GP or a general psychiatric outpatient unit prior to the study intervention. Other treatments are permitted for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Five Self-harm Behaviour Groupings Measure (5S-HM) | Treatment start, 3,6,9 and at end of treatment and at follow up at 24 months.
  Indirect and direct self-harm

SECONDARY OUTCOMES:
The World Health Organization Disability Assessment Schedule II (WHODAS 2) | Treatment start, 3,6,9 and at end of treatment and at follow up at 24 months.
  Daily functioning and impairment
The Borderline Symptom List-23 (BSL-23) | Treatment start, 3,6,9 and at end of treatment and at follow up at 24 months.
  Borderline symptoms
The Level of Personality Functioning Scale-Brief Form 2.0 (LPFS 2.0) | Treatment start, 3,6,9 and at end of treatment and at follow up at 24 months.
  Personality functioning
The Personality Inventory for DSM-V Brief Form (PID-5-BF) | Treatment start, 3,6,9 and at end of treatment and at follow up at 24 months.
  Personality structure
Hospitilization days | Treatment at end of treatment and at follow up at 24 months.
  Days admitted to a psychiatric ward past year

CONTACTS AND LOCATIONS:
Locations (1):
- Lund adult psychiatric hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Possibly not aoolicable due to Swedish data protection law

REFERENCES:
- [Background] Alvarez-Tomas I, Ruiz J, Guilera G, Bados A. Long-term clinical and functional course of borderline personality disorder: A meta-analysis of prospective studies. Eur Psychiatry. 2019 Feb;56:75-83. doi: 10.1016/j.eurpsy.2018.10.010. Epub 2018 Dec 24. PMID 30599336
- [Background] van Asselt AD, Dirksen CD, Arntz A, Severens JL. The cost of borderline personality disorder: societal cost of illness in BPD-patients. Eur Psychiatry. 2007 Sep;22(6):354-61. doi: 10.1016/j.eurpsy.2007.04.001. Epub 2007 Jun 4. PMID 17544636
- [Background] Chen SY, Cheng Y, Zhao WW, Zhang YH. Effects of dialectical behaviour therapy on reducing self-harming behaviours and negative emotions in patients with borderline personality disorder: A meta-analysis. J Psychiatr Ment Health Nurs. 2021 Dec;28(6):1128-1139. doi: 10.1111/jpm.12797. Epub 2021 Sep 20. PMID 34519138
- [Background] Cipriano A, Cella S, Cotrufo P. Nonsuicidal Self-injury: A Systematic Review. Front Psychol. 2017 Nov 8;8:1946. doi: 10.3389/fpsyg.2017.01946. eCollection 2017. PMID 29167651
- [Background] Ellison WD, Rosenstein LK, Morgan TA, Zimmerman M. Community and Clinical Epidemiology of Borderline Personality Disorder. Psychiatr Clin North Am. 2018 Dec;41(4):561-573. doi: 10.1016/j.psc.2018.07.008. Epub 2018 Oct 16. PMID 30447724
- [Background] Gad MA, Pucker HE, Hein KE, Temes CM, Frankenburg FR, Fitzmaurice GM, Zanarini MC. Facets of identity disturbance reported by patients with borderline personality disorder and personality-disordered comparison subjects over 20 years of prospective follow-up. Psychiatry Res. 2019 Jan;271:76-82. doi: 10.1016/j.psychres.2018.11.020. Epub 2018 Nov 10. PMID 30469092
- [Background] Gratz KL, Bardeen JR, Levy R, Dixon-Gordon KL, Tull MT. Mechanisms of change in an emotion regulation group therapy for deliberate self-harm among women with borderline personality disorder. Behav Res Ther. 2015 Feb;65:29-35. doi: 10.1016/j.brat.2014.12.005. Epub 2014 Dec 13. PMID 25557395
- [Background] Weekers LC, Hutsebaut J, Kamphuis JH. The Level of Personality Functioning Scale-Brief Form 2.0: Update of a brief instrument for assessing level of personality functioning. Personal Ment Health. 2019 Feb;13(1):3-14. doi: 10.1002/pmh.1434. Epub 2018 Sep 19. PMID 30230242
- [Background] Kaufman EA, Meddaoui B. Identity pathology and borderline personality disorder: an empirical overview. Curr Opin Psychol. 2021 Feb;37:82-88. doi: 10.1016/j.copsyc.2020.08.015. Epub 2020 Aug 25. PMID 32932110
- [Background] Krueger RF, Derringer J, Markon KE, Watson D, Skodol AE. Initial construction of a maladaptive personality trait model and inventory for DSM-5. Psychol Med. 2012 Sep;42(9):1879-90. doi: 10.1017/S0033291711002674. Epub 2011 Dec 8. PMID 22153017
- [Background] Kroger C, Harbeck S, Armbrust M, Kliem S. Effectiveness, response, and dropout of dialectical behavior therapy for borderline personality disorder in an inpatient setting. Behav Res Ther. 2013 Aug;51(8):411-6. doi: 10.1016/j.brat.2013.04.008. Epub 2013 May 14. PMID 23727659
- [Background] Mehlum L. Mechanisms of change in dialectical behaviour therapy for people with borderline personality disorder. Curr Opin Psychol. 2021 Feb;37:89-93. doi: 10.1016/j.copsyc.2020.08.017. Epub 2020 Aug 25. PMID 32979766
- [Background] McMain SF, Fitzpatrick S, Boritz T, Barnhart R, Links P, Streiner DL. Outcome Trajectories and Prognostic Factors for Suicide and Self-Harm Behaviors in Patients With Borderline Personality Disorder Following One Year of Outpatient Psychotherapy. J Pers Disord. 2018 Aug;32(4):497-512. doi: 10.1521/pedi_2017_31_309. Epub 2017 Sep 14. PMID 28910214
- [Background] Meuldijk D, McCarthy A, Bourke ME, Grenyer BF. The value of psychological treatment for borderline personality disorder: Systematic review and cost offset analysis of economic evaluations. PLoS One. 2017 Mar 1;12(3):e0171592. doi: 10.1371/journal.pone.0171592. eCollection 2017. PMID 28249032
- [Background] Schmitgen MM, Niedtfeld I, Schmitt R, Mancke F, Winter D, Schmahl C, Herpertz SC. Individualized treatment response prediction of dialectical behavior therapy for borderline personality disorder using multimodal magnetic resonance imaging. Brain Behav. 2019 Sep;9(9):e01384. doi: 10.1002/brb3.1384. Epub 2019 Aug 14. PMID 31414575
- [Background] Levi FA, Hrushesky WJ, Blomquist CH, Lakatua DJ, Haus E, Halberg F, Kennedy BJ. Reduction of cis-diamminedichloroplatinum nephrotoxicity in rats by optimal circadian drug timing. Cancer Res. 1982 Mar;42(3):950-5. PMID 7199382
- [Background] Woodbridge J, Reis S, Townsend ML, Hobby L, Grenyer BFS. Searching in the dark: Shining a light on some predictors of non-response to psychotherapy for borderline personality disorder. PLoS One. 2021 Jul 27;16(7):e0255055. doi: 10.1371/journal.pone.0255055. eCollection 2021. PMID 34314461